CLINICAL TRIAL: NCT06899971
Title: The Association Between Tau & GFAP and Postoperative Neurological Impairment in Patients Undergoing Cardiac Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, Principal Investigator, MD, Boston Children's Hospital
Other Study IDs: IRB-P00050907
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery Requiring Cardiopulmonary Bypass; Brain Injury; Congenital Heart Defect
MeSH Terms: conditions — Brain Injuries; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Patients less than 18 years old who undergo cardiac surgical procedures on cardiopulmonary bypass.
  Interventions: Other: Collecting discarded blood samples

INTERVENTIONS:
Other: Collecting discarded blood samples — Discarded blood samples will be collected from routine clinical labs collected before and after surgery.

SUMMARY:
Patients born with heart defects often undergo surgical procedures on a heart lung machine. With improvements in medical and surgical management, their survival has significantly improved, but their brain insult has not been paid much attention. This study is to determine the relationship between specific proteins in the blood and brain injury in patients less than 18-year-old undergoing heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* less than 18 years old
* undergoing cardiac surgery with cardiopulmonary bypass at Boston Children's Hospital

Exclusion Criteria:

* undergoing an emergent procedure and do not have more than 1 hour ahead of time to review the consent
* patient in a moribund condition American Society of Anesthesiology (ASA 5)
* patient with a hematological and/or oncological disease
* Jehovah witnesses
* patient on preoperative mechanical ventilation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients less than 18 years old undergoing a cardiac surgical procedure at Boston Children's Hospital with cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of postoperative neurological impairment | 24 hours following surgery
  Understand the correlation between measured proinflammatory cytokines and several proteins that are highly expressed in brain cells with postoperative neurological status.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States